CLINICAL TRIAL: NCT03420248
Title: Comparison of Pain After Uterine Artery Embolization Using Non-spherical Polyvinyl Alcohol Particles or Tris-acryl Gelatin Microsphere in Patients With Symptomatic Fibroids
Brief Title: Comparison of Pain of Two Different Methods in Uterine Artery Embolization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Assistant professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2016-1108
Record Dates: First submitted 2018-01-16; First posted 2018-02-05 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Leiomyoma
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-spherical polyvinyl alcohol particle (Experimental): For embolic material, non-spherical polyvinyl alcohol particle is used.
  Interventions: Device: Non-spherical polyvinyl alcohol particle or Tris-acryl gelatin microsphere
- Tris-acryl gelatin microsphere (Experimental): For embolic material, Tris-acryl gelatin microsphere is used.
  Interventions: Device: Non-spherical polyvinyl alcohol particle or Tris-acryl gelatin microsphere

INTERVENTIONS:
Device: Non-spherical polyvinyl alcohol particle or Tris-acryl gelatin microsphere — One of non-spherical polyvinyl alcohol particle or tris-acryl gelatin microsphere is used for embolic materials. All other processes are same.

SUMMARY:
The primary purpose of this study is to compare pain after uterine artery embolization using non-spherical polyvinyl alcohol particles or tris-acryl gelatin microsphere in patients with symptomatic fibroids

DETAILED DESCRIPTION:
Uterine artery embolization(UAE) is a minimally invasive treatment alternative to hysterectomy and myomectomy in symptomatic fibroids. However, post-procedural pain after UAE remains a major problem. The non-spherical polyvinyl alcohol particle and tri-acryl gelatin microsphere are two embolic materials used for UAE.Therefore, the aim of study is to compare pain intensity and inflammation after uterine artery embolization using non-spherical polyvinyl alcohol particles or tris-acryl gelatin microsphere in patients with symptomatic fibroids

ELIGIBILITY:
Inclusion Criteria:

* Uterine artery embolization due to multiple fibroids

Exclusion Criteria:

* Severe liver or kidney dysfunction
* Drug allergy
* Bradycardia (<45 bpm) or heart block
* Uncontrolled hypertension

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity by numerical rating scale | 0-24 h after UAE
  0-10 numerical rating scale (0, no pain at all; 10, worst pain imaginable

SECONDARY OUTCOMES:
C-reactive protein | 24 h after UAE
  mg/L
White blood cell count | 24 h after UAE
  /uL
Neutrophil percentage | 24 h after UAE
Neutrophil-to-lymphocyte ratio | 24 h after UAE
Platelet-to-lymphocyte ratio | 24 h after UAE
Mean platelet volume | 24 h after UAE
  fL(femtolitre)
Sucessful rate at 3 month after UAE measured by MRI | 3 month after UAE
  Complete necrosis incidence

CONTACTS AND LOCATIONS:
Overall Officials: So Yeon Kim, MD, PhD, Principal Investigator — Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Severance Hospital, Yonsei University College of Medicine; Man Deuk Kim, MD, PhD, Principal Investigator — Department of Radiology, Research Institute of Radiological Science, Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Sesverance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No